CLINICAL TRIAL: NCT07189663
Title: Study on the Correlation Between Serum and Fecal Sialic Acid Levels and Tumor Characteristics as Well as Postoperative Anastomotic Leakage in Patients With Colorectal Tumors
Status: Not yet recruiting | Type: Observational
Sponsor: Xiaolong Li (Other)
Responsible Party: Sponsor-Investigator, Xiaolong Li, Investigator, Army Medical University, China
Organization: Army Medical University, China (Other)
Other Study IDs: 2025-study268-02; 2019R68 (Other Grant/Funding Number: ArmyMedChina)
Record Dates: First submitted 2025-09-22; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Neoplasia; Anastomotic Leakage
Keywords: colorectal neoplasia; anastomotic leakage; sialic acid
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Fecal samples (5-7g) were collected routinely for intestinal flora analysis (16SrRNA sequencing). Fecal samples were collected and stored immediately at-80 ° C for subsequent DNA extraction.(1) Fecal sialic acid testing: high performance liquid chromatography (HPLC) testing prospectively collected
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Serum Sialic Acid (SA) High-Level Group: For the Retrospective Section , record the serum sialic acid (SA) levels of enrolled subjects. Using the median of these levels as the cutoff, assign patients with levels above the median to Serum Sialic Acid (SA) High-Level Group
- Serum Sialic Acid (SA) Low-Level Group: For the Retrospective Section , record the serum sialic acid (SA) levels of enrolled subjects. Using the median of these levels as the cutoff, assign patients with levels under the median to Serum Sialic Acid (SA) Low-Level Group
- Fecal Sialic Acid (SA) High-Level Group: For the prospective Section , record the fecal sialic acid (SA) levels of enrolled subjects. Using the median of these levels as the cutoff, assign patients with levels above the median to Fecal Sialic Acid (SA) High-Level Group
- Fecal Sialic Acid (SA) Low-Level Group: For thr prospective Section , record the fecal sialic acid (SA) levels of enrolled subjects. Using the median of these levels as the cutoff, assign patients with levels under the median to Fecal Sialic Acid (SA) Low-Level Group

SUMMARY:
This is a Single-center bidirectional cohort study combined with prospective sample analysis conducted by the Department of General Surgery at the Second Affiliated Hospital of Army Medical University (Xinqiao Hospital).

The purpose of this study was to retrospectively collect the preoperative serum sialic acid content and postoperative pathological data of colorectal cancer patients in our hospital's medical order system (including tumor size and stage, etc.) and anastomotic leakage, and analyze the correlation between serum sialic acid content and pathological characteristics of tumor and the correlation between anastomotic leakage; and further collect the feces of colorectal cancer patients in our hospital for 16S microbiome sequencing, and detect their sialic acid content, and observe the relationship between fecal sialic acid content and tumor size and stage; Intestinal flora composition and postoperative anastomotic leakage correlation, provide a new theoretical basis for the prevention and treatment of postoperative anastomotic malhealing.

DETAILED DESCRIPTION:
Background#Colorectal cancer (CRC) is one of the most common gastrointestinal malignancies worldwide, ranking third in incidence and second in mortality among all cancers. Surgical resection remains the primary treatment for CRC, particularly for early- and mid-stage patients, as it effectively removes tumor tissue and prolongs survival. However, postoperative anastomotic healing failure (e.g., anastomotic leakage) is a severe complication of colorectal surgery, with an incidence rate of 5%-20%. Anastomotic leakage not only significantly increases postoperative mortality but also prolongs hospital stays, escalates medical costs, and imposes a heavy burden on both patients and healthcare systems. The pathogenesis of anastomotic leakage is complex,involving factors such as local ischemia, surgical technique, infection, and gut microbiota dysbiosis. In recent years, with advancements in microbiomics research, the role of gut microbiota in anastomotic healing has gained increasing attention.

During malignant transformation, colorectal cancer cells exhibit significantly upregulated expression of sialic acid (SA) on their cell surfaces. Sialic acid, a class of nine-carbon monosaccharides widely distributed on mammalian cell surfaces, participates in cell-cell recognition, immune regulation, and host-microbe interactions. Studies have shown that shed sialic acid from colorectal tumor cells enters the intestinal lumen, serving as a critical nutrient source for gut microbes. Notably, certain pathogens (e.g., Escherichia coli, Klebsiella pneumoniae) can utilize sialic acid as a carbon source to promote their proliferation and colonization. These pathogens may impair anastomotic healing through multiple mechanisms: first, by disrupting the intestinal mucosal barrier and exacerbating local inflammation; second, by inhibiting epithelial cell repair and delaying tissue regeneration; and third, by producing toxins or metabolites that further damage local tissues. Thus, colorectal tumor-derived sialic acid may indirectly increase the risk of postoperative anastomotic healing failure by nourishing specific pathogens. Although existing research suggests that sialic acid from colorectal tumors influences the gut microenvironment by feeding pathogens, the specific mechanisms underlying its impact on postoperative anastomotic healing remain unclear. This hypothesis requires experimental validation.

The purpose of this study was to retrospectively collect the preoperative serum sialic acid content and postoperative pathological data of colorectal cancer patients in our hospital's medical order system (including tumor size and stage, etc.) and anastomotic leakage, and analyze the correlation between serum sialic acid content and pathological characteristics of tumor and the correlation between anastomotic leakage; and further collect the feces of colorectal cancer patients in our hospital for 16S microbiome sequencing, and detect their sialic acid content, and observe the relationship between fecal sialic acid content and tumor size and stage; Intestinal flora composition and postoperative anastomotic leakage correlation, provide a new theoretical basis for the prevention and treatment of postoperative anastomotic malhealing.

Study Design# This study was carried out in the general surgery department of our hospital. Based on the hospital electronic medical record system (EMR), the data of patients meeting the standard from January 2010 to December 2020 were retrospectively extracted, and the stool samples and clinical data of patients scheduled for surgery from August 2025 to August 2026 were prospectively collected.

Primary Objective:Anastomotic fistula occurrence, changes in flora structure Key Outcomes# Data Analysis: Data extracted from electronic medical records. Statistical analysis using SPSS 22.0 (χ² test for categorical data, t-test for normally distributed continuous data; significance p<0.05). Ethics: Approved by the institutional ethics committee. Conducted in accordance with the Declaration of Helsinki and Chinese regulations. Patient privacy and data confidentiality are prioritized. Timeline: Patient data collection and analysis (Aug 2025-Aug 2026); Statistical analysis and manuscript preparation (Sep-Dec 2025). Significance:The purpose of this study was to retrospectively collect the preoperative serum sialic acid content and postoperative pathological data of colorectal cancer patients in our hospital's medical order system (including tumor size and stage, etc.) and anastomotic leakage, and analyze the correlation between serum sialic acid content and pathological characteristics of tumor and the correlation between anastomotic leakage; and further collect the feces of colorectal cancer patients in our hospital for 16S microbiome sequencing, and detect their sialic acid content, and observe the relationship between fecal sialic acid content and tumor size and stage; Intestinal flora composition and postoperative anastomotic leakage correlation, provide a new theoretical basis for the prevention and treatment of postoperative anastomotic malhealing.

ELIGIBILITY:
Inclusion Criteria: For the retrospective Part : Age between 18 and 80 years; Patients who underwent radical resection of colorectal cancer in our hospital from January 2010 to December 2020; Preoperative serum sialic acid level was measured (a routine test item in liver function biochemical tests in our hospital from 2010 to 2020); Complete postoperative pathological data.

* For the prospective Section:Age between 18 and 80 years; Patients who underwent radical resection of colorectal cancer in our hospital from August 2025 to August 2026; Voluntarily sign the informed consent form for fecal sample collection.

Exclusion Criteria:

* Emergency surgery, palliative surgery, or concurrent other malignant tumors; Preoperative neoadjuvant chemoradiotherapy (may affect SA levels and microbiota); Recent infection: history of severe infection within 3 months before surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent radical resection of colorectal cancer in the Department of General Surgery, Xinqiao Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1468 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2026-09-10 (Estimated); Study Completion 2026-11-10 (Estimated)

PRIMARY OUTCOMES:
The occurrence of anastomotic fistula | From enrollment to the end of treatment at 1 month
  This study will statistically analyze the occurrence of anastomotic fistula in postoperative patients and explore its risk factors

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Army Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
We are currently planning to conduct a series of studies. As data sharing will be postponed until all studies have been completed, the data will not be made available at this time